CLINICAL TRIAL: NCT04207008
Title: iBDecide Pilot Randomized Controlled Trial
Brief Title: Trial of a Decision Support Intervention for Adolescents and Young Adults With Ulcerative Colitis
Acronym: iBDecide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Ellen A. Lipstein MD, MPH, Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-1103a
Record Dates: First submitted 2019-12-11; First posted 2019-12-20 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Ulcerative Colitis, Pediatric
Keywords: Adolescents and young adults; decision making
MeSH Terms: conditions — Pediatric ulcerative colitis

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iBDecide App Decision-support Arm (Experimental): Participants will download the iBDecide app on their smartphone approximately two weeks prior to the scheduled clinic visit. Approximately one week after the clinic visit, survey data, along with demographic data will be collected from all participants via a brief telephone call. We will collect data on app use between installation and the clinic visit as well as in the 3 months following the clinic visit.
  Interventions: Other: iBDecide Decision Support Application
- Control Arm (No Intervention): Control participants will not use the iBDecide app prior to their clinic visit. They will complete a brief telephone survey approximately one week from clinic visit.

INTERVENTIONS:
Other: iBDecide Decision Support Application — The iBDecide app provides an electronic tools to learn more about UC, track symptoms, create a nutrition diary, enter reminders for medication and clinic visits, as well as learn more about treatment options and compare UC medications.
  Arms: iBDecide App Decision-support Arm

SUMMARY:
A web application decision support tool has been developed for adolescents and young adults (AYAs). The purpose of this pilot trial is to test the web application for adolescent and young adults (AYAs) with Ulcerative Colitis (UC). This research will assess acceptability, feasibility of the decision support intervention for AYA UC patients. Participants will be randomized to usual care or usual care plus the web application prior to an upcoming clinic visit in Gastroenterology. Participants will complete surveys one week after their clinic visit about decision making preferences and, for those in the intervention group, usability and acceptability of the web application.

DETAILED DESCRIPTION:
The iBDecide app provides participants with electronic tools to learn more about UC, track symptoms, create a nutrition diary, enter reminders for medication and clinic visits, as well as learn more about treatment options and compare UC medications.

Participants will be provided instructions over the phone or via email to download the iBDecide app on their personal smartphone approximately two weeks prior to the scheduled clinic visit. When possible they will download the app during the consent call and the research staff member will review features of the app with the participant. For those unable to download it while talking on the phone, a follow-up phone call will be scheduled to review the features. During the consenting phone call or at the clinic visit, a time will be scheduled to collect additional information via a brief telephone survey approximately one week after the clinic visit. Participants will be sent emails and an electronic calendar invitation to confirm their scheduled telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients with Ulcerative Colitis that have an appointment at the CCHMC Gastroenterology clinic
* 14-25 years of age
* Treatment decision anticipated during clinic
* Did not participate in usability testing for the iBDecide App
* Has a smart phone that can download the iBDecide app

Exclusion Criteria:

* Unable to read or speak English

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | At clinic visit
  The extent to which this intervention impacts the flow of a clinic appointment, as measured by physician perception of visit length and efficiency.
Acceptability of intervention | One week after clinic visit
  The extent to which patients and physicians feel the intervention is appropriate and useful. This is measured through adaptations of the System Usability Scale and the decision aid acceptability measure.

SECONDARY OUTCOMES:
Decisional conflict | At clinic visit
  Measure of decisional uncertainty, assessed via Decisional Conflict Scale.
Perceived Shared Decision making | One week after clinic visit
  Degree of shared decision-making the patient and physician each report, measured by the Shared Decision-Making Questionnaire-9 and Shared Decision-making Questionnaire 9-doc.
Decision preference congruence | One week after clinic visit
  Extent to which the patients' role in the decision process matched their preferred role, measured via the Control Preference Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Lipstein, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matula KA, Minar P, Daraiseh NM, Lin L, Recker M, Lipstein EA. Pilot trial of iBDecide: Evaluating an online tool to facilitate shared decision making for adolescents and young adults with ulcerative colitis. Health Expect. 2022 Dec;25(6):3105-3113. doi: 10.1111/hex.13618. Epub 2022 Sep 26. PMID 36161973